CLINICAL TRIAL: NCT06580405
Title: A Feasibility Study to Evaluate the Safety of the KNP-1000 Apheresis System in Patients With Preeclampsia With Severe Features
Brief Title: A Feasibility Study to Evaluate the Safety of the KNP-1000 Apheresis System in Severe Preeclampsia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kaneka Medical America LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KNP-1000-US01
Record Dates: First submitted 2024-08-23; First posted 2024-08-30 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Pre-Eclampsia, Severe
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- KNP-1000 Apheresis System (Experimental): Participants are to be treated with the system up to 2 times per week, continuing through delivery or 34 weeks of pregnancy, whichever comes first.
  Interventions: Device: KNP-1000 Apheresis System

INTERVENTIONS:
Device: KNP-1000 Apheresis System — sFlt-1 is removed from the participants' plasma through treatment.

SUMMARY:
The study will primarily evaluate safety of the KNP-1000 apheresis system for pregnant women and their fetuses diagnosed with preeclampsia with severe features between 23- and 32-weeks' gestation (very preterm).

ELIGIBILITY:
Inclusion Criteria:

A participant is deemed suitable for inclusion in the investigation if she meets the following criteria:

1. Pregnant woman ≥ 23 0/7 and < 32 0/7 weeks gestation, aged 18 to 45 years, hospitalized for preeclampsia at time of enrollment.
2. Severe hypertension ever defined by resting systolic BP ≥ 160 mm Hg and/or diastolic BP ≥ 110 mm Hg on two occasions measured at least 4 hours apart.
3. Proteinuria, defined as ≥ 300 mg protein in a 24-hour urine collection or ≥ 0.3 protein/creatinine ratio.
4. Provision of signed and dated informed consent form.

Exclusion Criteria:

A participant will be excluded from the investigation if any of the following maternal or fetal criteria are met.

Maternal Exclusion Criteria:

1. Documented history of chronic hypertension, defined as systolic BP ≥ 140mmHg and/or systolic BP ≥ 90 mmHg before pregnancy or prior to 20 weeks of gestation.
2. Documented history of proteinuria prior to pregnancy or prior to 20 weeks of gestation.
3. Taking any form of angiotensin cascade blocker or angiotensin-converting enzyme (ACE) inhibitor at time of enrollment.
4. Documented history of cardiac impairments including uncontrolled arrhythmia, unstable angina, decompensated congestive heart failure, or valvular disease.
5. Actively receiving therapeutic anticoagulation therapy or within the therapeutic window after ceasing anticoagulation therapy at the time of enrollment.
6. Any condition which, in the opinion of the Investigator, would necessitate immediate delivery within 24 hours.
7. Signs or history of cerebral nervous system dysfunction, including seizures, cerebral edema (previously confirmed by computed tomography scan or magnetic resonance imaging per medical records).
8. Confirmed or suspected diagnosis of pulmonary edema at time of enrollment.
9. Diagnosis of HELLP syndrome.
10. Thrombocytopenia (platelet count < 100,000/mm3) at time of enrollment.
11. Anemia defined as hemoglobin < 8 g/dL at time of enrollment.
12. Absent or reverse flow on umbilical Doppler ultrasound exam at the time of screening, or documented history of negative or reverse flow during the current gestation period.
13. Diagnosis of placenta previa during the current gestation period.
14. Preterm labor at or before time of screening.
15. Documented medical history of active hepatitis B virus, hepatitis C virus (HCV), syphilis, tuberculosis infection, or human immunodeficiency virus (HIV) positive status.
16. Any condition that the Investigator deems a risk to the study participant or fetus in completing the investigation.
17. Hypersensitivity to dextran sulfate cellulose or heparin.
18. Multiple gestation.
19. Documented history of familial hypercholesterolemia.
20. Suspicion or diagnosis of placental abruption during the current gestation.
21. Patients who have received the drug treatment not recommended by the American College of Obstetricians and Gynecologists (ACOG) practice bulletin Gestational Hypertension and Preeclampsia (the clinical management guidelines) within 6 months prior to enrollment.
22. Patients who have participated in another clinical trial within 6 months prior to enrollment.

Fetal Exclusion Criteria:

1. Documented record of chromosomal anomalies.
2. Identifiable structural fetal abnormalities present at time of screening or a record of such abnormalities prior to enrollment.
3. Oligohydramnios, defined as Amniotic fluid index (AFI) less than 5 cm when measured using the four-quadrant method at time of enrollment.
4. Fetal growth restriction (FGR) defined as estimated fetal weight (EFW) below the 5th percentile for gestational age.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Estimated)
Dates: Start 2025-05-31 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Antepartum maternal and fetal device-related serious adverse events | Until date of delivery
  Rate of antepartum maternal and fetal device-related serious adverse events
Postpartum maternal and neonatal device-related serious adverse events | Following delivery until end of follow-up (2 years)
  Rate of postpartum maternal and neonatal device-related serious adverse events
Maternal, fetal, and neonatal mortality | Until end of follow-up (2 years)
  Rate of maternal, fetal, and neonatal mortality
Obstetric complication | Until discharge or 6 weeks after delivery, whichever occurs first
  Incidence rate of obstetric complication
Fetal complications | Until date of delivery
  Incidence rate of fetal complications
Neonatal morbidities associated with premature delivery | Following delivery until discharge or 6 weeks after delivery, whichever occurs first
  Incidence rate of neonatal morbidities associated with premature delivery
Neonatal intensive care unit (NICU) admissions | From date of NICU admission until the date of NICU discharge, assessed up to 24 months
  Rate of NICU admissions and length of stay

SECONDARY OUTCOMES:
Prolongation of pregnancy | Until date of delivery
  Number of days from enrollment to delivery
Maternal systolic blood pressure | Until discharge or 6 weeks after delivery, whichever occurs first
  Change in maternal systolic blood pressure over the duration of the investigation
Maternal diastolic blood pressure | Until discharge or 6 weeks after delivery, whichever occurs first
  Change in maternal diastolic blood pressure over the duration of the investigation
Maternal proteinuria | Until discharge or 6 weeks after delivery, whichever occurs first, an average of 4 months
  Change in maternal proteinuria before and after each procedure
Gestational age of the neonate at delivery | At date of delivery
  Gestational age of the neonate at delivery
Weight of neonate at delivery | At date of delivery
  Weight of neonate at delivery
Amniotic fluid volume | Until the date of delivery, an average of 3 months
  Change in amniotic fluid volume before and after each procedure
Fetal umbilical artery flow | Until the date of delivery, an average of 3 months
  Change in fetal umbilical artery flow before and after each procedure
Uterine artery flow | Until the date of delivery, an average of 3 months
  Change in uterine artery flow before and after each procedure
Maternal low-density lipoprotein cholesterol (LDL-C) levels | Until discharge or 6 weeks after delivery, whichever occurs first, an average of 4 months
  Change in LDL-C levels in maternal serum before and after each procedure
Fetal growth restriction | Until date of delivery
  Incidence rate of fetal growth restriction
APGAR scores | At date of delivery
  Neonatal APGAR scores
Umbilical artery and vein blood gases | At date of delivery
  Umbilical artery and vein blood gases
Bayley Scales | At 6, 12, and 24 months after delivery
  Bayley Scales of Infant and Toddler Development, Fourth Edition assessment at 6, 12, and 24 months after delivery. Standard score (Composite score) range from 40 to 160, with higher scores indicating higher performance.
Body weight of infant | Following delivery until end of follow-up (2 years)
  Body weight (grams) of infant at birth and during extended follow-up
Body length and head circumference of infant | Following delivery until end of follow-up (2 years)
  Body length and head circumference (centimeters) of infant at birth and during extended follow-up

OTHER OUTCOMES:
Soluble fms-like tyrosine kinase-1 (sFlt-1)/ placental growth factor (PlGF) ratio in maternal serum | Until discharge or 6 weeks after delivery, whichever occurs first
  sFlt-1/PlGF ratio in maternal serum
Percentage reduction of sFlt-1 levels in maternal serum | Until the date of delivery, an average of 3 months
  Percentage reduction of sFlt-1 levels in maternal serum after each apheresis treatment
Change in sFLT-1 levels | During each apheresis procedure
  Change in sFLT-1 levels between the inlet and outlet of the apheresis system
Change in PlGF levels | During each apheresis procedure
  Change in PlGF levels between the inlet and outlet of the apheresis system